CLINICAL TRIAL: NCT06388460
Title: Asthma Link: A Partnership Between Pediatric Practices, Schools, and Families to Improve Medication Adherence and Health Outcomes in Children With Poorly Controlled Asthma
Brief Title: Asthma Link Effectiveness Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Trivedi, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001015; R01HL169229 (NIH)
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Childhood Asthma
Keywords: asthma; childhood asthma; medication adherence; school-supervised asthma therapy; real-world
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asthma Link (Experimental): Practices in the Asthma Link condition will receive brief training on how to identify, refer and arrange for children with poorly controlled asthma to receive school-supervised therapy with the child's school health staff. Participants will receive an educational asthma workbook.
  Interventions: Other: Asthma Link
- Enhanced Usual Care (Active Comparator): Practices in the Enhanced Usual Care condition will receive brief training on how to identify and refer the same group of children with poorly controlled asthma and these children will receive an educational asthma workbook.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Asthma Link — Providers enroll patients to receive school-supervised asthma therapy and an asthma educational workbook
  Arms: Asthma Link
Other: Enhanced Usual Care — Providers enroll patients to receive an asthma educational workbook
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this cluster Randomized Control Trial is to determine the effectiveness of Asthma Link, a school supervised asthma therapy program, compared with an educational asthma workbook, in improving asthma symptoms for children with poorly controlled asthma aged 5-14.

DETAILED DESCRIPTION:
Asthma is an extremely common chronic disease in childhood with significant morbidity. The majority of asthma morbidity in children is due to medication non-adherence, and both morbidity and medication non-adherence disproportionately impact minoritized children. School-supervised asthma therapy ensures that children receive their preventive asthma medication daily at school and has shown efficacy in improving medication adherence and asthma health outcomes, particularly in low-income and racial/ethnic minority children. However, this strategy has not been widely adopted in practice to produce meaningful public health impact. To address this gap, the study team developed a new model, Asthma Link, which partners pediatric practices, schools, and families to deliver school-supervised asthma therapy. This intervention leverages established infrastructure and requires minimal resources to operate, enhancing sustainability in a real-world setting. The pilot trial of Asthma Link showed improved asthma symptoms when compared to an enhanced usual care condition, particularly among low-income, Black and Latino children, and demonstrated trial feasibility. Moreover, the research team has rigorously adapted this intervention for real-world use using input from diverse, multi-level community stakeholders.

This 14 site cluster randomized controlled trial will determine the effectiveness of Asthma Link versus an enhanced usual care condition in improving asthma health outcomes in school-aged children with poorly controlled asthma.

The investigators central hypothesis is that children in Asthma Link will have higher Asthma Control Test scores at 6 months compared with children in enhanced usual care; with maintained improvements at 12 months. The secondary hypothesis is that children in Asthma Link will have higher inhaled corticosteroid adherence and quality of life scores, and lower rates of asthma exacerbations, school absences and parental lost workdays compared with children in the enhanced usual care condition.

ELIGIBILITY:
STUDY INCLUSION/EXCLUSION CRITERIA:

Child Inclusion Criteria:

* Meet the eligibility criteria for Asthma Link (as described below)
* Enrolled in Asthma Link (if randomized to the Asthma Link Condition)
* Able and willing to provide informed assent

Child Exclusion Criteria:

* Unable or unwilling to provide informed assent
* Developmental delay that would prevent study participation.

Parent Inclusion Criteria:

* Parent/guardian to patient
* 18 years or older
* Able to understand and communicate in English or Spanish
* Able and willing to provide informed consent.

Child eligibility for children enrolled in Asthma Link:

* children aged 5-14 years (enrolled in grade K-8)
* prescribed daily inhaled corticosteroid (ICS) for asthma
* Asthma Control Test (ACT) score ≤19 OR 1 or more of ANY of following in the past 1 year: course of oral steroids, hospitalization, Emergency Department visit, sick visit for asthma
* parent/child report of poor ICS adherence on adherence checklist- i.e. child or parent says "Yes" when provider asks if they have difficulty remembering to take their medication or if they regularly take medication holidays or breaks
* able and willing to assent
* parental permission
* English or Spanish speaking

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Improving Asthma Symptoms | Baseline, 6 months, 12 months
  Asthma Control Test to measure child's asthma control on a scale of 0-25. A score of 19 or less is considered poorly controlled asthma.

SECONDARY OUTCOMES:
Improving Medication Adherence | Baseline, 6 months, 12 months
  Survey to measure medication adherence
Improving Healthcare Utilization | Baseline, 6 months, 12 months
  Survey questions to measure # of emergency room visits, # of hospital admissions, # of oral steroid courses due to asthma
Reducing Parental Lost Workdays | Baseline, 6 months, 12 months
  Survey to measure the number of days a parent has missed work
Reducing School Absences | Baseline, 6 months, 12 months
  Survey to measure the number of days a child has missed school
Improving Quality of Life | Baseline, 6 months, 12 months
  Survey to measure the quality of life of the child and parent

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Trivedi, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No